CLINICAL TRIAL: NCT03845335
Title: Clinical Performance Evaluation of a Hyaluronic Acid-coated Hybrid Dental Implant Compared to a Non-Coated Standard Rough Dental Implant: A Pragmatic Multi-center Randomized Controlled Trial
Brief Title: Clinical Performance Evaluation of Two Different Dental Implants
Acronym: HAHy-vs-C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Elite Odontoiatrica (Other)
Responsible Party: Principal Investigator, Luca Ferrantino, Researcher, Elite Odontoiatrica
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol 01
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Edentulism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both patients and clinicians will be unaware of treatment allocation until the randomization sequence is disclosed. Clinician who will perform test and control treatment will know the group allocation.
  Clinician who will do the outcome evaluation will be unaware of the treatment allocation.
  A blinded researcher will perform data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HA-coated hybrid implant (Experimental): Patient allocated to this group will receive an iMAX® Hyaluronic Acid-coated hybrid dental implant for their dental implant-supported restoration.
  Interventions: Device: dental implant-supported restoration
- Moderately rough implant (Active Comparator): Patient allocated in this group will receive an iMAX® non-coated moderately rough dental implant with a machined neck their dental implant-supported restoration.
  Interventions: Device: dental implant-supported restoration

INTERVENTIONS:
Device: dental implant-supported restoration — During the oral surgery session for dental implant insertion, after implant site preparation, the opaque sealed envelope containing the patient allocation will be opened. Following the group allocation, the patient will receive either an HA-coated Hybrid or moderately rough dental implant

SUMMARY:
In brief, the aim of this randomized controlled trial is to evaluate the patient satisfaction and the clinical performance of two types of implants: 1) HA-coated hybrid dental implant and 2) non-coated moderately rough dental implant. The comparison will be studied during a routine implant placement of experienced dental implantologists.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate to the present investigation
* Psychological appropriateness and good compliance to dentist instructions
* Patient who have been selected for implant therapy by an experienced surgeon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Survival Rate | 12 months after implant placement
  Cumulative implant survival rate

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Elite Odontoiatrica Magenta, Magenta, MI
  - Elite Odontoiatrica Milano, Milan, MI
  - Elite Odontoiatrica Opera, Opera, MI
  - Elite Odontoiatrica Caronno, Caronno Pertusella, VA

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] de Bruyn H, Collaert B, Linden U, Bjorn AL. Patient's opinion and treatment outcome of fixed rehabilitation on Branemark implants. A 3-year follow-up study in private dental practices. Clin Oral Implants Res. 1997 Aug;8(4):265-71. doi: 10.1034/j.1600-0501.1997.080403.x. PMID 9586472
- [Background] Jung RE, Pjetursson BE, Glauser R, Zembic A, Zwahlen M, Lang NP. A systematic review of the 5-year survival and complication rates of implant-supported single crowns. Clin Oral Implants Res. 2008 Feb;19(2):119-30. doi: 10.1111/j.1600-0501.2007.01453.x. Epub 2007 Dec 7. PMID 18067597
- [Background] Lang NP, Zitzmann NU; Working Group 3 of the VIII European Workshop on Periodontology. Clinical research in implant dentistry: evaluation of implant-supported restorations, aesthetic and patient-reported outcomes. J Clin Periodontol. 2012 Feb;39 Suppl 12:133-8. doi: 10.1111/j.1600-051X.2011.01842.x. PMID 22533953
- [Background] Meijndert L, Meijer HJ, Stellingsma K, Stegenga B, Raghoebar GM. Evaluation of aesthetics of implant-supported single-tooth replacements using different bone augmentation procedures: a prospective randomized clinical study. Clin Oral Implants Res. 2007 Dec;18(6):715-9. doi: 10.1111/j.1600-0501.2007.01415.x. Epub 2007 Sep 20. PMID 17888016
- [Background] Pjetursson BE, Tan K, Lang NP, Bragger U, Egger M, Zwahlen M. A systematic review of the survival and complication rates of fixed partial dentures (FPDs) after an observation period of at least 5 years. Clin Oral Implants Res. 2004 Dec;15(6):625-42. doi: 10.1111/j.1600-0501.2004.01117.x. PMID 15533124
- [Background] Pjetursson BE, Tan WC, Zwahlen M, Lang NP. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. J Clin Periodontol. 2008 Sep;35(8 Suppl):216-40. doi: 10.1111/j.1600-051X.2008.01272.x. PMID 18724852